CLINICAL TRIAL: NCT05588596
Title: Developing and Validating an Integrative Model Incorporating Mindfulness-based Resilience Intervention to Address Post-Traumatic Stress Disorder in People Living With HIV
Brief Title: Intervention Program to Address PTSD in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, TANG Chulei, Principal investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018040
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: HIV; AIDS; Mindfulness-based Stress Reduction; China; Resilience; PTSD
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Access to routine hospital care and outpatient services. Patients received relevant health counseling provided by the investigator. In addition, Patients received Trauma Resiliency Mindfulness-Informed Intervention, including Mindfulness awareness, body scanning, walking awareness, mindful breathing, etc.
  Interventions: Behavioral: Trauma Resiliency Mindfulness-Informed Intervention
- Waitlist group (No Intervention): Access to routine hospital care and outpatient services. In addition, the patient received relevant health counseling provided by the investigator, including AIDS related knowledge counseling, diet advice, etc. At the end of the study, patients in the waitlist group were provided with intervention.

INTERVENTIONS:
Behavioral: Trauma Resiliency Mindfulness-Informed Intervention — The total duration of the intervention was once a week for eight weeks. The aim of the intervention was to teach patients a range of trauma recovery mindfulness skills
  Arms: Intervention group

SUMMARY:
The goal of this randomised controlled trial is to evaluate the efficacy of an integrated intervention program on post-traumatic stress disorder (PTSD) symptoms and related physiological and psychological indicators of people living with HIV (PLWH). The main question it aims to answer are:

* to evaluate the efficacy of the intervention program on PTSD symptoms and related physiological and psychological indicators of PLWH through empirical research.
* to analyze the mechanism of the intervention. Eligible PLWH were recruited and randomly divided as intervention group and control group. The efficacy of Trauma Resiliency Mindfulness-Informed Intervention on PTSD symptoms and related physiological and psychological indicators in PLWH was evaluated at baseline, after intervention, and 3 months after intervention through this randomized controlled trial.

Researchers compared the intervention group and control group to see if it was feasible and had potential clinical value to introduce the Trauma Resiliency Mindfulness-Informed intervention program into the management of PLWH in China.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* been diagnosed with HIV for more than 1 month
* screened positive with PTSD CheckList - Civilian Version (PCL-C)
* voluntary participation

Exclusion Criteria:

* impaired Verbal Communication
* have received psychological treatment or related psychological intervention in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Change of PTSD symptoms | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  PTSD CheckList - Civilian Version (PCL-C) was used. The scale consists of 17 items divided into 3 dimensions. Each dimension is scored from 1 to 5. The total score of PCL-C ranges from 17 to 85, with higher scores indicating severer PTSD symptoms.

SECONDARY OUTCOMES:
Change of depression symptoms | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  The Zung Self-Rating Depression Scale (SDS) was used. The scale consists of 20 items. Each dimension is scored from 1 to 4. The total score ranges from 20 to 80, with higher scores indicating severer depression symptoms.
Change of resilience | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  The Connor-Davidson Resilience Scale (CD-RISC) was used. The scale consists of 25 items. Each dimension is scored from 0 to 4. The total score ranges from 0 to 100, with higher scores indicating higher resilience.
Change of rumination | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  The Ruminative Responses Scale (RRS) was used. The scale consists of 22 items. Each dimension is scored from 1 to 4. The total score ranges from 22 to 88, with higher scores indicating higher rumination
Change of perceived social support | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  The Multidimensional Scale of Perceived Social Support (MSPSS) was used. The scale consists of 12 items. Each dimension is scored from 1 to 7. The total score ranges from 12 to 84, with higher scores indicating higher perceived social support.
Change of mindfulness | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  The Short Inventory of Mindfulness Capability (SIM-C) was used. The scale consists of 12 items. Each dimension is scored from 1 to 5. The total score ranges from 12 to 60, with higher scores indicating higher mindfulness.

OTHER OUTCOMES:
Change of medication adherence | Outcomes were evaluated at baseline, immediately after the intervention, and 3 months follow-up after the intervention
  0 (0%)~10 (100%) grade was adopted for scoring. Evaluate the condition of patients taking antiretroviral drugs according to doctor's orders in the past month

CONTACTS AND LOCATIONS:
Overall Officials: Chulei TANG, Doctor, Principal Investigator — Central South University
Locations (1):
- The First Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF